CLINICAL TRIAL: NCT04614766
Title: A Phase 1/2 Trial Using AZEDRA and LUTATHERA in a Dosimetrically-determined Optimal Combination for Therapy of Selected Patients With Midgut Neuroendocrine Tumors
Brief Title: A Clinical Trial Evaluating the Safety of Combining Lutathera(R) and Azedra(R) to Treat Mid-gut Neuroendocrine Tumors
Acronym: SPORE-3
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Azedra withdrawn from US market
Sponsor: David Bushnell (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David Bushnell, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202005556; P50CA174521 (NIH)
Record Dates: First submitted 2020-10-13; First posted 2020-11-04 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Gastro-enteropancreatic Neuroendocrine Tumor; Neuroendocrine Tumors
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate; 3-Iodobenzylguanidine

STUDY DESIGN:
Intervention Model Description: Participants who do not meet eligibility criteria for the combined therapy will be asked to participate in the active comparator, which is single agent Lutathera administered as per FDA guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination Therapy (Experimental): Combined treatment with Lutathera® and Azedra® Administered amounts of each drug are based on imaging and radiation dose constraints to the kidneys and the bone marrow. The drug administration is individualized to each participant.
  Interventions: Drug: Lutathera; Drug: Azedra
- Lutathera® only (Active Comparator): Single agent Lutathera® administered per standard of care: 200 millicuries of drug every 8 weeks for a total of 4 doses.
  Interventions: Drug: Lutathera

INTERVENTIONS:
Drug: Lutathera — intravenous administration
  Other Names: lutetium Lu 177 dotatate
Drug: Azedra — intravenous administration
  Other Names: iobenguane I-131
  Arms: Combination Therapy

SUMMARY:
This study is designed to identify the best tolerated doses of Lutathera® and Azedra® when co-administered to treat midgut neuroendocrine tumors. These drugs are radioactive drugs, known as radionuclide therapy, and are both approved in the treatment of midgut neuroendocrine tumor as single agents (not together). Currently, the safest and best tolerated doses of these drugs (when combined) is unknown. That is the purpose of this clinical trial.

DETAILED DESCRIPTION:
Azedra and Lutatheraare are FDA-approved radioactive drugs designed to treat specific tumor cells. These drugs are a combination of the radiation (131-Iodine, 177-lutetium) and a protein that targets the tumor cell (MIBG or DOTATATE). Because these proteins are attracted to, and stick to, the tumor, the radiation is centered in the tumors. This kills more tumor cells and minimizes radiation-damage to healthy tissues, like the heart and lungs.

Two organs still absorb some of the radiation, though: bone marrow and the kidney. These organs limit how much radiation can be given to tumors, but we don't know how much radiation is too much. Too much radiation to bone marrow can result in anemia. Too much radiation to the kidneys can result in kidney failure. From prior radiation therapies, we have a general idea of how much radiation we can give safely.

Azedra and Lutathera have never been given together. We want to give them together because many times, tumors are actually groups of different types of cells. This means, not all the cells respond to therapy the same way. If some tumor cells survive therapy, the tumor will continue to grow and eventually come back. We know some mid-gut neuroendocrine tumors (NETs) have targets for DOTATATE and some other mid-gut NETs have targets for MIBG. We also have now identified that some people with mid-gut NETs have different tumors: some with targets for MIBG and some with targets for DOTATATE. For these people, this means treating only with Azedra or Lutathera will not be enough to treat their cancer. They need both radioactive drugs.

Because we are combining these radioactive drugs, this study is known as a first-in-man study. We are also using a special imaging to help us estimate the radiation dose to the bone marrow and to the kidneys. This is what decides the final dose of Azedra and Lutathera.

After receiving a standard treatment of Lutathera, participants are asked to undergo imaging to verify they have both MIBG and DOTATATE tumor types:

* participants are given a tracer dose of Azedra
* a special camera (SPECT/CT) collects images (scans)
* imaging (scans) are done over 4 calendar days
* blood samples are taken at that time, too, to measure the circulating amount of tracer doses

If the scans show a participant does not have both MIBG and DOTATATE receptors, they continue with standard therapy (Lutathera only). Participants are asked to still undergo study assessments to provide a comparison group.

If the scans show a participant has both MIBG and DOTATATE receptors, combined therapy is administered:

* a customized dose of Lutathera is given on day 1 of a treatment cycle. This is given outpatient.
* a customized dose of Azedra is given on day 2 of a treatment cycle. This is given inpatient (admitted to the hospital).
* participants are monitored through blood tests to identify the side effects of therapy.

Each participant can have up to 2 cycles of therapy. The cycles are 12 weeks apart.

The doses for Lutathera and Azedra are decided based on radiation to the bone marrow and radiation to the kidney. Doses are decided by how well other participants have done on this study.

Participants have life long follow-up for this study. This is very important, because a study like this has not been done.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to provide informed consent; legally authorized representative will not be utilized compliant with the principles of good clinical practice (i.e., ICH E6(R2)).
* Stated willingness to comply with all study procedures and availability for duration of study
* Aged ≥ 18 years to 80 years at the time of study drug administration
* Pathologically confirmed (histology or cytology) malignant neoplasm that is determined to be:

  * a well-differentiated neuroendocrine tumor (i.e. grade 1 or grade 2) with a primary tumor location believed to be midgut, or,
  * pheochromocytoma, or,
  * paraganglioma
* Recommended to receive LUTATHERA® or AZEDRA® therapy
* Disease measuring ≥ 1.5 cm in diameter on CT or MRI as measured per RECIST
* Adequate performance status (ECOG of 0 or 1; or KPS of >70).
* Agrees to contraception during therapy.
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patient with increased fall risk in the opinion of healthcare professionals
* Women who are pregnant.
* Women who are breast feeding.
* Surgery, radiation therapy, or chemotherapy ≤ 4 weeks of C1D1. (Toxicities from prior therapies should have resolved to ≤ CTCAE grade 1 or a new baseline established).
* Prior peptide-receptor radiotherapy (PRRT).
* Therapeutic investigational drug within 4 weeks of C1D1 (imaging agents are acceptable).
* A concurrent malignancy that, in the opinion of the investigator, would cause a safety risk by delaying therapy or confound/negatively impact study objectives (documentation of the rationale must be provided).
* History of congestive heart failure with a history of cardiac ejection fraction ≤ 35%.
* Patients unable to discontinue medications known to affect MIBG uptake (unless approved by the PI or designee)
* Proteinuria grade 2 (i.e., 2+ proteinuria).
* Prior external beam radiation dose of >16 Gy to the kidneys.
* Prior external beam radiation (including brachytherapy) involving 25% of the bone marrow (excluding scatter doses of 5 Gy) as estimated by a radiation oncologist.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Octreoscan® or Netspot™.

Participants meeting the above criteria will receive one cycle of standard Lutathera treatment (200 millicuries) as well as a tracer dose of Azedra for imaging. Participants will then undergo protocol specific imaging to calculate the radiation dose to the kidneys, the bone marrow, and to the tumor lesions.

To continue on study and receive the combined therapy, a participant's imaging must demonstrate one of the following:

* At least one tumor that is positive for Azedra but negative for Lutathera in addition to Lutathera positive tumors, or,
* At least one tumor site where the calculated safe radiation dose to that tumor site is 25% higher using the combined therapy compared to Lutathera alone

Participants who do not meet this criteria are invited to participate in the comparator arm to receive standard Lutathera treatment as indicated by their physicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Phase 1: Determination of maximum tolerated radiation dose (MTD) to the kidneys | 9 months after initial treatment
  MTD will be determined by incidence of renal AEs as characterized by type, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study therapy.
Phase 1: Determination of maximum tolerated radiation dose (MTD) to the bone marrow. | 9 months
  MTD will be determined by incidence of hematologic AEs as characterized by type, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study therapy.
Phase 2: Objective Response Rate (ORR) | 6 months post-treatment
  Objective response rate, measured using standardized RECIST criteria, is a reflection of complete tumor response and partial tumor response when obtained at 6 months and 12 months post-treatment.
Phase 2: Objective Response Rate (ORR) | 12 months post-treatment
  Objective response rate, measured using standardized RECIST criteria, is a reflection of complete tumor response and partial tumor response when obtained at 6 months and 12 months post-treatment.

SECONDARY OUTCOMES:
Tumor size | 6 months post-treatment
  Determine tumor size and response using RECIST 1.1 criteria in patients treated with the combined regimen
Tumor size | 12 months post-treatment
  Determine tumor size and response using RECIST 1.1 criteria in patients treated with the combined regimen
Number of Treatment-Related Adverse Events | Up to 24 months post-treatment
  Categorize and quantify adverse events using the Common Terminology Criteria for Adverse Events (v5)

CONTACTS AND LOCATIONS:
Overall Officials: David Bushnell, M.D., Principal Investigator — The University of Iowa and the Iowa City VAMC
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants must opt in to data sharing. For those that do, imaging, adverse event, and treatment data will be provided.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: phase 1 data: 12 months after identifying the maximum dose phase 2 data: 12 months after last participant last visit
Access Criteria: A data usage agreement and privacy contract will need to be completed between investigators and their institutions. Data are to be destroyed after completion / use.

REFERENCES:
- [Background] Madsen MT, Bushnell DL, Juweid ME, Menda Y, O'Dorisio MS, O'Dorisio T, Besse IM. Potential increased tumor-dose delivery with combined 131I-MIBG and 90Y-DOTATOC treatment in neuroendocrine tumors: a theoretic model. J Nucl Med. 2006 Apr;47(4):660-7. PMID 16595501
- [Background] Bushnell DL, Madsen MT, O'cdorisio T, Menda Y, Muzahir S, Ryan R, O'dorisio MS. Feasibility and advantage of adding (131)I-MIBG to (90)Y-DOTATOC for treatment of patients with advanced stage neuroendocrine tumors. EJNMMI Res. 2014 Dec;4(1):38. doi: 10.1186/s13550-014-0038-2. Epub 2014 Sep 10. PMID 26116109